CLINICAL TRIAL: NCT02307240
Title: Phase I Open Label, Multi-center Study to Assess the Safety, Tolerability and Pharmacokinetics of Orally Administered CUDC-907, an HDAC and PI3K Inhibitor, in Subjects With Advanced/Relapsed Solid Tumors
Brief Title: Open Label, Multi-center Study to Assess the Safety, Tolerability and Pharmacokinetics of CUDC-907 in Subjects With Advanced/Relapsed Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-907-102
Record Dates: First submitted 2014-11-18; First posted 2014-12-04 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Triple-Negative Breast Cancer; High-grade Serous Ovarian Cancer; Solid Tumors; NUT Midline Carcinoma
Keywords: TNBC; HGSOC; NMC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — CUDC-907

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CUDC-907 - five days on/two days off (Experimental): 60 mg/day CUDC-907, oral administration, five days on/two days off until disease progression or other discontinuation criteria are met.
  Interventions: Drug: CUDC-907

INTERVENTIONS:
Drug: CUDC-907 — CUDC-907 oral with meals.

SUMMARY:
This is a Phase I, open-label, multi-center trial designed to evaluate the safety, tolerability and pharmacokinetics of CUDC-907 administered orally to subjects with advanced/relapsed solid tumors.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multi-center trial designed to evaluate the safety, tolerability and pharmacokinetics of CUDC-907 administered orally to subjects with advanced/relapsed solid tumors. The following dosing schedule, consisting of 21-day treatment cycles, is being examined:

Five days on/two days off on Days 1 to 5, 8 to 12, and 15 to 19 (5/2 schedule).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age for solid tumor; in the case of midline carcinoma with NUT rearrangement. subjects may be ≥16 years of age.
2. Histopathologically confirmed diagnosis of an advanced solid tumor such as breast cancer or midline carcinoma with NUT rearrangement, that has progressed despite standard therapy, or for which no standard therapy exists. For enrollment in the expansion cohorts, histopathological confirmation of triple-negative breast cancer or high-grade serous ovarian cancer is required.
3. Measurable or evaluable disease.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Recovery to Grade 1 or baseline of any toxicity due to prior systemic treatments or radiotherapy (excluding alopecia).

Exclusion Criteria:

1. Systemic anticancer therapy within three weeks of study entry, except for nitrosoureas or mitomycin C within six weeks.
2. Radiotherapy within one week prior to starting study treatment.
3. Other investigational agent(s) within 21 days prior starting to study treatment.
4. Symptomatic central nervous system (CNS) involvement or lymphangitic metastasis. Stable or improving CNS disease that is not under active treatment after receipt of adequate therapy is allowed.
5. Uncontrolled or severe cardiovascular disease, including myocardial infarction or unstable angina within six months prior to study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease or cardiac amyloidosis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-11; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of oral CUDC-907 in subjects with advanced/relapsed solid tumors | 21 day cycle

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of CUDC-907; Pharmacokinetic parameters will include area under the concentration-time curve (AUC). | 21 day cycle
To evaluate biomarkers of CUDC-907 activity | 24 months
To assess the preliminary anti-cancer activity of CUDC-907 | 24 months
  The Investigator will evaluate each subject for response to therapy according to standard response criteria for each individual subject's tumor type

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCSF School of Medicine, San Francisco, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas